CLINICAL TRIAL: NCT00176033
Title: Influence of Drug Transporter Expression on the Pharmacokinetics of the HIV Protease Inhibitor Kaletra (Lopinavir/Ritonavir) and on the Concentration Relations Between Plasma, Blood Cells, Saliva and Urine
Brief Title: Influence of Drug Transporter Expression on the Pharmacokinetics of the HIV Protease Inhibitor Kaletra
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: K026
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Healthy; Pharmacokinetics
Keywords: ritonavir; lopinavir; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aim of this study is to determine the pharmacokinetics of Kaletra™ (HIV protease inhibitors lopinavir and ritonavir) in different body compartments and to assess the role of four different drug transporters (MDR, MRP1, MRP2 and BCRP) in the tissue distribution of the two protease inhibitors. The latter will be studied by comparing intracellular concentrations of peripheral blood mononuclear cells (PBMCs) with total and free plasma concentrations in healthy individuals. These effects will be studied after single dose (day 1), during steady state (day 3), and during chronic treatment (day 14).

DETAILED DESCRIPTION:
Objective:

Measurement of AUC, Cmax, tmax, t1/2 and clearance (Cl) of the protease inhibitor Kaletra™ (lopinavir and ritonavir) each in the plasma of healthy individuals

* establish free and total plasma - blood cell concentration-relationship
* establish free and total plasma - saliva concentration-relationship
* establish blood cell concentration - drug transporter expression-relationship

ELIGIBILITY:
Inclusion Criteria:

* Good state of health

Exclusion Criteria:

* Drug treatment with known inhibitors or inducers of cytochrome P450 isozymes or ABC-transporters within the preceding 2 months
* Any acute or chronic illness
* Smoking
* Pregnancy
* Alcohol or drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, MD, BSc, Principal Investigator — Department of Internal Medicine VI
Locations (1):
- Clinical Research Center, Department of Internal Medicine VI, Heidelberg, Germany